CLINICAL TRIAL: NCT00713765
Title: A Double-blind, Randomised, Cross-over, Placebo-controlled Study of Repeated Oral Doses of AZD3480 and a Single Dose of Donepezil to Evaluate the Pharmacokinetic Interaction Between AZD3480 and Donepezil in Healthy Extensive and Poor Metabolisers of CYP2D6
Brief Title: Pharmacokinetic Interaction Between AZD3480 and Donepezil
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Ended prematurely - The trial never commenced.
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: D3690C00005; EudraCt No.2008-002847-17
Record Dates: First submitted 2008-07-09; First posted 2008-07-11 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-08

CONDITIONS: Alzheimer's Disease
Keywords: Healthy volunteers
MeSH Terms: conditions — Alzheimer Disease | interventions — ispronicline; Donepezil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): AZD3480 + Donepezil
  Interventions: Drug: AZD3480; Drug: Donepezil

INTERVENTIONS:
Drug: AZD3480 — 18 total doses of 40 mg, on days 1-18
Drug: Donepezil — One single dose of mg on day 5

SUMMARY:
The aims of this study are to 1) examine the effects of AZD3480 and donepezil on the blood concentrations of each other and 2) assess the safety and tolerability of the combined administration of AZD3480 with donepezil.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study-specific procedures
* BMI between 18 and 30 kg/m2
* Medical and surgical history and physical examination without any clinically significant findings
* Genotyped as an EM, defined in this study as having ≥ 1.5 functional CYP2D6 alleles, or a PM, defined as having zero functional CYP2D6 alleles

Exclusion Criteria:

* History of clinically significant cardio- or cerebrovascular, pulmonary, renal, hepatic, neurological, mental or gastrointestinal disorder or any other major disorder that may interfere with the objectives of the study, as judged by the Investigator
* Clinically significant illness as judged by the Investigator, within two weeks before the first administration of investigational product
* Female subjects who have a positive pregnancy test or who are pregnant or breast-feeding

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2008-12; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
PK variables | Frequent sampling occasions during

SECONDARY OUTCOMES:
Safety variables (adverse events, blood pressure, pulse, safety lab) | During the whole treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Hans Göran Hårdemark, Study Director — AstraZeneca R&D, Sodertalje, Sweden; Simon Constable, Principal Investigator — ICON Development Solutions, Manchester, UK
Locations (1):
- Research Site, Manchester, United Kingdom

REFERENCES:
- See also: D3690C00005_No_Results_Certificate — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1367&filename=D3690C00005.pdf